CLINICAL TRIAL: NCT00510224
Title: A Phase II Study of the Somatostatin Analog Sandostatin LAR in Patients With Androgen Independent Prostate Cancer
Brief Title: Sandostatin for Patients With Androgen Independent Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped at interim analyses phase due to lack of efficacy
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF055514
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sandostatin

INTERVENTIONS:
Drug: Sandostatin — Sandostatin 30mg intramuscular every 28 days

SUMMARY:
This is an open label, single center Phase II trial of Sandostatin LAR in patients with hormone refractory prostate cancer. Patients will receive Sandostatin LAR 30 mg intramuscularly every 28 days. Patients will be treated until the time of disease progression, unacceptable toxicity or withdrawal of consent. The study will require 27 evaluable patients.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate changes in prostate specific antigen (PSA) in patients with androgen independent prostate cancer who are treated with Sandostatin LAR.

Secondary Objective:

To evaluate the effects of Sandostatin LAR on circulating levels of Insulin Growth Factor-1 and Insulin Growth Factor Binding Protein 1.

To evaluate the safety of Sandostatin LAR in this patient population. To evaluate the pre versus post treatment mitogenic effects of serum derived from subjects with prostate cancer compared to pretreatment serum.

Patients with androgen independent prostate cancer who do not have bone or visceral metastases are selected for this trial because they are a patient population that is likely to have no symptoms from the disease or rapid progression that would suggest the need for chemotherapy. Additionally, given the preclinical data suggesting that IGF-1 expression and signaling occurs concomitantly with the onset of androgen independent growth, it is felt that testing in the "early" androgen independent state is warranted. This trial is consistent with overall goal to develop IGF-1 targeted therapies in patients with disease progression and a lower disease burden.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Biochemical disease progression following androgen deprivation and therapy with at least one antiandrogen defined as three rises in PSA with PSA determinations at least 4 weeks apart and each PSA value > 0.2 ng/ml.
* Four weeks since prior therapy with Flutamide.
* Six weeks since prior therapy with Bicalutamide or Nilutamide.
* Current PSA > 5 ng/ml.
* Testosterone <50 ng/dL.
* SGPT (ALT) < 1.5 times upper limit of normal.
* Fasting blood glucose > 60 mg/dL.
* ECOG performance status 0, 1 or 2.
* No visceral or bony metastatic disease (Lymph node only metastases are allowed).
* No prior chemotherapy for prostate cancer.
* No current treatment with insulin or an oral hypoglycemic.
* No history of treatment with octreotide analogs for prostate cancer.
* No NYHA Class 3 or 4 cardiac status.

Exclusion Criteria:

* Diabetes Mellitus requiring medical therapy and/or that which is not controlled by dietary means (HbA1C<6.0).
* A history of gallstones that has been clinically significant. Patients who have undergone cholecystectomy are eligible.
* Other concomitant medical or psychiatric condition which would make it undesirable, in the physician's opinion, for the patient to participate in the protocol or would jeopardize compliance with the protocol requirements.
* Prior treatment with chemotherapy for prostate cancer.
* No current treatment with Saw Palmetto, or Proscar. Patients must be off these medicines for more than 4 weeks.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Friedlander TW, Weinberg VK, Small EJ, Sharib J, Harzstark AL, Lin AM, Fong L, Ryan CJ. Effect of the somatostatin analog octreotide acetate on circulating insulin-like growth factor-1 and related peptides in patients with non-metastatic castration-resistant prostate cancer: results of a phase II study. Urol Oncol. 2012 Jul-Aug;30(4):408-14. doi: 10.1016/j.urolonc.2010.06.014. Epub 2010 Oct 2. PMID 20884247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men with prostate adenocarcinoma that had progressed despite androgen deprivation therapy were recruited for participation at one U.S. clinical site (UCSF)
Groups:
- Octreotide Acetate: Octreotide acetate 30mg intramuscular every 28 days
Period: Overall Study
Arm/Group | Octreotide Acetate
Started | 13
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Octreotide Acetate
Number analyzed (Participants) | 13
Age Continuous [Median (Full Range); unit: years] | 75 [63 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 13
Primary therapy [Number; unit: participants] — Type of therapy prior to study enrollment
  participants
    Prostatectomy | 3
    Radiation Therapy | 6
    Androgen Deprivation | 4
Median PSA [Median (Full Range); unit: ng/ml] — PSA was measured by chemiluminescent immunoassay on the Immulite 2000 analyzer (Siemens Healthcare Diagnostics, Deerfield, IL)
  ng/ml | 36.2 [5.4 to 342.8]
Gleason Score [Median (Full Range); unit: Score] — A Gleason score is assigned by a pathologist based on the sum of two numbers: the first number is the grade of the most common tumor pattern, the second number is the grade of the second most common pattern. For example, if the most common tumor pattern was grade 3, but some cells were found to be grade 4, the Gleason Score would be 3+4 = 7. The Gleason Score ranges from 2 to 10, with 10 having the worst prognosis.
  Score | 8 [5 to 10]
Hemoglobin [Median (Full Range); unit: gm/dl] | 13.9 [9.5 to 16.5]

OUTCOME MEASURES:

1. Primary Outcome: PSA Response
Description: Number of participants with a PSA decline of at least 50% from Baseline during the first 3 cycles of therapy, confirmed by a second measurement at least 2 weeks later.
Time Frame: 12 weeks
Population: n=27 was determined to be sufficient to test for a 20% PSA response proportion compared with a null hypothesis of 5%. A two-stage design was employed to carry out an interim analysis for efficacy. As no patient showed a PSA decline among the first 13 accrued after 3 cycles (the first evaluation of PSA response), accrual was discontinued
Measure: Number; unit: Participants
Arm/Group | Octreotide Acetate
Number analyzed (Participants) | 13
Participants | 0

2. Secondary Outcome: Pre-post Percent Change in Circulating Levels of IGF-1 and IGF-Binding Protein 1.
Description: Serum was batched and IGF and IGFBP levels were assayed at one time at the end of the study using an enzyme-linked immunoabsorbent assay (ELISA) method by Diagnostic Systems Laboratories (Webster, TX).
Time Frame: Baseline, 12 weeks
Measure: Median (Full Range); unit: percent change
Arm/Group | Octreotide Acetate
Number analyzed (Participants) | 13
percent change
  IGF-1 | -34.5 [-57.4 to 11.1]
  IGFBP-1 | 76.3 [-45.1 to 589.6]

3. Secondary Outcome: Grade 4-5 Adverse Events
Time Frame: 12 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Octreotide Acetate
Number analyzed (Participants) | 13
Adverse Events | 0

4. Secondary Outcome: Pre Versus Post Treatment Mitogenic Effects.
Time Frame: 12 Weeks
Population: The trial was closed for futility after no PSA responses were observed among the first 13 patients, and this analysis was not performed
Arm/Group | Octreotide Acetate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: While on study therapy (9-51 weeks)
Arm/Group | Octreotide Acetate
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide Acetate (N=13)
Angina (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Elevated INR (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Headache (General disorders) | 1
Hepatic congestion (Hepatobiliary disorders) | 1
Hyperkalemia (Renal and urinary disorders) | 1
Pain (General disorders) | 1
Scleral hemorrhage (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes